CLINICAL TRIAL: NCT05028946
Title: A Phase IB Multiple Ascending Dose Study of Safety and Tolerability of Orally Administered Foralumab, a Fully Human Anti-CD3 Monoclonal Antibody, in Subjects With Moderate to Severely Active Crohn's Disease
Brief Title: A Study of Oral Foralumab in Participants With Moderate to Severely Active Crohn's Disease
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: For business reasons
Sponsor: Tiziana Life Sciences LTD (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: TILS-014; 2021-002698-24 (EudraCT Number)
Record Dates: First submitted 2021-08-24; First posted 2021-08-31 (Actual); Last update posted 2022-10-20 (Actual); Status verified 2022-10

CONDITIONS: Crohn's Disease
Keywords: Anti-CD3 Monoclonal Antibody; Inflammatory bowel disease; Oral anti-CD3
MeSH Terms: conditions — Crohn Disease; Inflammatory Bowel Diseases | interventions — foralumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Cohort 1: Foralumab Dose Level 1 (Experimental): Participants will receive foralumab enteric coated capsules at dose level 1, administered orally once daily for 2 weeks (5 consecutive days in each week with a 2-day undosed safety assessment period after each 5 day treatment period).
  Interventions: Drug: Foralumab
- Cohort 2: Foralumab Dose Level 2 (Experimental): Participants will receive foralumab enteric coated capsules at dose level 2, administered orally once daily for 2 weeks (5 consecutive days in each week with a 2-day undosed safety assessment period after each 5 day treatment period).
  Interventions: Drug: Foralumab
- Cohort 3: Foralumab Dose Level 3 (Experimental): Participants will receive foralumab enteric coated capsules at dose level 3, administered orally once daily for 2 weeks (5 consecutive days in each week with a 2-day undosed safety assessment period after each 5 day treatment period).
  Interventions: Drug: Foralumab
- Cohort 4: Foralumab Dose Level 4 (Experimental): Participants will receive foralumab enteric coated capsules at dose level 4, administered orally once daily for 2 weeks (5 consecutive days in each week with a 2-day undosed safety assessment period after each 5 day treatment period).
  Interventions: Drug: Foralumab

INTERVENTIONS:
Drug: Foralumab — Foralumab will be administered per dose and schedule specified in the arm description.
  Other Names: Human anti-CD3 monoclonal antibody (mAb)

SUMMARY:
The primary objective of this study is to establish the safety and tolerability of multiple ascending doses (MAD) of foralumab enteric coated capsules administered orally, once daily for 5 days per week over 2 weeks in participants with moderate to severely active Crohn's Disease (CD).

DETAILED DESCRIPTION:
Four different doses of foralumab enteric coated capsules will be studied for safety and tolerability in a MAD format. Participants in the sequential MAD cohorts will receive treatment when the safety data of one cohort are reviewed by the Data Safety Monitoring Board (DSMB) and are deemed favorable to proceed with the next treatment in the subsequent cohort.

ELIGIBILITY:
Inclusion Criteria:

* Participant has been diagnosed with active CD as confirmed by endoscopic examination with histological confirmation for at least 12 weeks before the screening visit; only study participant who has endoscopic examination by colonoscopy of disease location that includes ileocolon and/or colon and who has a Simple Endoscopic Score for Crohn's Disease (SES-CD) ≥3 will be enrolled in the study.
* Participant has a CDAI ≥220 but ≤450 points (that is, participant has moderate to severely active disease despite current treatment).
* Participant is naïve to anti-CD3 therapy.
* Non-smoker or use of nicotine or other nicotine-containing products (snuff, chewing tobacco, cigars, pipes, e-cigarettes or nicotine-replacement products such as nicotine chewing gum and nicotine plasters) will not be allowed from 3 months before the screening visit until the final follow-up visit.
* Participant's current regimen of concomitant medication(s) falls within the definitions provided in the protocol.
* Participant must weigh ≥50 kg at the time of signing informed consent.
* Male or female

  1. Sexually active male participant must agree to use highly effective contraception as detailed in of this protocol during the treatment period and for at least 10 weeks after the last dose of study medication (or longer if required by local approved label).
  2. A female participant is eligible to participate if she is not pregnant, not breastfeeding, and at least one of the following conditions applies:

  i) Not a woman of childbearing potential (WOCBP). ii) A WOCBP who agrees to follow the guidance for highly effective contraception during the treatment period and for at least 10 weeks after the last dose of study medication (or longer if required by local approved label).

Exclusion Criteria:

* Participant has symptomatic coronavirus disease of 2019 (COVID-19) or a positive severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) test result prior to screening.
* Participant has a suspected or confirmed diagnosis of ulcerative colitis (UC), indeterminate colitis, ischemic colitis, radiation colitis, diverticular disease associated with colitis, or microscopic colitis.
* Participant with any known fistula involving the gastrointestinal (GI) tract (except for perianal fistula).
* Participant with symptomatic stricturing type disease at the time of the screening visit.
* Participant has had an extensive colonic resection, subtotal or total colectomy, diagnosis of short bowel syndrome or a history of >3 small bowel resections.
* Participant has a functional colostomy or ileostomy. Exception: A participant who has had a temporary stoma in the past, which has been reversed, may be enrolled.
* Participant has had a surgical bowel resection within 6 months before the screening visit or is planning any resection at a time while enrolled in the study.
* Participant with clinical suspicion of intra-abdominal abscess(es). If a participant receives treatment for the abscess, they may be rescreened.
* Participant currently requires or is anticipated to require surgical intervention for CD during the study.
* Participant has a current or recent history (within 6 months before the screening visit) of clinically relevant renal, hepatic, hematological, GI (other than CD), endocrine, pulmonary, neurological, or cerebral disease including blood dyscrasia (for example, pancytopenia, aplastic anemia), demyelinating disease (for example, multiple sclerosis, myelitis, optic neuritis), or ischemic heart disease.
* Participant has known history of or current clinically active infection with histoplasma, coccidioides, paracoccidioides, pneumocystis, tuberculous mycobacteria, nontuberculous mycobacteria, blastomyces, aspergillus, legionella, or listeria.
* Participant with evidence of an acquired or congenital immunodeficiency state, including, but not limited to, known human immunodeficiency virus (HIV) infection, agammaglobulinemia, organ transplantation, T cell deficiencies, or human T cell lymphotropic virus type 1.
* Participant has a history of chronic or recurrent infections (more than 3 episodes requiring antibiotics/antivirals during the preceding year), recent serious or life-threatening infection within the 4 weeks prior to the screening visit (including Herpes zoster), infection requiring intravenous (IV) antibiotic use within the 4 weeks prior to the screening visit or oral antibiotic use within the 2 weeks prior to the screening visit.
* Participant has a concurrent malignancy or a history of any malignancy at any time (including nonmelanoma skin cancer).
* Participant has concurrent bowel dysplasia or a history of bowel dysplasia in the 5 years before the screening visit.
* Participant has a history of a lymphoproliferative disorder, including lymphoma, or signs and symptoms suggestive of lymphoproliferative disease at any time.
* Participant has a known hypersensitivity to any excipients of the investigational medicinal product (IMP) or its ingredients.
* Participant is currently receiving chronic concomitant systemic antibiotic therapy for diseases other than CD or acne.
* Participant received any live (includes attenuated) vaccination within the 10 weeks prior to the screening visit or intending to receive during the study (inactivated vaccinations are permitted at any time prior to and during the study) or within 3 months after last dose of certolizumab pegol (CZP) or foralumab.
* Participant has a positive fecal laboratory test result for enteric pathogens and/or ova and parasites at the screening visit.
* Participant who has evidence of, or treatment for clostridium difficile infection or other intestinal pathogen, within 28 days prior to first dose of study medication.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-05-01 (Estimated); Primary Completion 2023-07-07 (Estimated); Study Completion 2023-11-07 (Estimated)

PRIMARY OUTCOMES:
Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs) | Day 1 up to Day 14
  Adverse events categorized and graded via CTCAE

SECONDARY OUTCOMES:
Change From Baseline in Crohn's Disease Activity Index (CDAI) Score at Day 5 and Day 12 | Baseline, Day 5 and Day 12
  The CDAI score is used to quantify the symptoms of participants with Crohn's Disease. CDAI scores generally range from 0 to 600 points. A score of 150 or below indicates remission and a score above 450 indicates extremely severe disease. A decrease in CDAI over time indicates improvement in disease activity.

IPD SHARING:
Plan to Share IPD: No